CLINICAL TRIAL: NCT04263571
Title: Hepcidin as a Predictor for the IVI Mediated Increase in Haemoglobin Levels Prior to Elective Surgery
Brief Title: Hepcidin as a Predictor for the IVI Mediated Increase in Haemoglobin Levels
Acronym: PREDICT-IVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Goethe University (Other)
Collaborators: Pharmacosmos A/S (Industry); University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Priv.-Doz. Dr. Andrea Ulrike Steinbicker, Prof. Dr. Andrea Ulrike Steinbicker, Goethe University
Other Study IDs: 06-AnIt-18
Record Dates: First submitted 2019-08-30; First posted 2020-02-11 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Anemia; IV Iron
Keywords: hemoglobin; hepcidin
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a multidisciplinary study, which involves all kind of medical specialties. Patients, who are scheduled for elective surgery, will be seen at a multidisciplinary anaesthesia/Patient Blood Management (PBM) clinic and screened for anaemia prior to surgery. Anaemic patients will eventually be treated with 500mg of iron isomaltoside.

DETAILED DESCRIPTION:
Hgb levels, standard iron parameters and hepcidin will be assessed. Additional parameters that might influence Hgb or IVI levels will be documented.

All main analyses will be pre-defined in detail in a statistical analysis plan. In order to analyse the responsiveness to IVI, the change in Hgb levels from PBM clinic to day 0 will be analysed using multivariable regression models. The association of change in Hgb and hepcidin will be analysed adjusting for potentially confounding factors as age, gender or number of days from PBM clinic to surgery. The correlation of hepcidin and standard iron parameters will be assessed. Based on the increase in Hgb levels, responders to IVI will be defined. The definition of good- bad responder in terms of delta Hgb levels depends on the time between IVI substitution and surgery. ROC analyses will be performed and potential predictors (e.g. hepcidin, ferritin) will be compared concerning the area under the ROC curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* iron deficiency anemia
* elective surgery planned during the next 4 to 28 days

Exclusion Criteria:

* Contraindications for an IV iron Infusion severe infections, hepatocellular carcinoma, liver metastases, acute severe asthma, a simultaneous oral iron medication, another IV iron preparation, iron overload, chronic renal failure and regular IV iron substitution
* Pregnancy or lactation
* Allergy against iron
* chronic renal failure on dialysis
* iron overload

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with iron deficiency anemia prior to elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic.
  Change in hemoglobin level after IV iron treatment

SECONDARY OUTCOMES:
Hepcidin | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic.
  Serum hepcidin level prior to IV iron Infusion (ng/ml)
Serum iron | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Serum iron prior to IV iron
Transferrin saturation | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Transferrin saturation prior to IV iron
Ferritin levels | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Ferritin levels prior to IV iron
Transferrin protein | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Transferrin protein prior to IV iron
Soluble transferrin receptor | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Soluble transferrin receptor prior to IV iron
Number of reticulocyte counts | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Number of reticulocyte counts
Mean corpuscular hemoglobin (MCH) | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Mean corpuscular hemoglobin prior to IV iron
Level of reticulocyte-Hb in g/dl | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Level of reticulocyte-Hb prior to IV iron
Level of Phosphate in serum | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Level of Phosphate in serum prior to IV iron
Corpuscular hemoglobin of reticulocytes (CHr) | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Value of each parameter prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Corpuscular hemoglobin of reticulocytes (CHr) prior to IV iron
Leucocyte count | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. value prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Leucocyte count prior to IV iron Infusion
Level of C-reactive Protein | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. value prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Level of C-reactive Protein prior to IV iron Infusion
Level of Serum Procalcitonin | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. value prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Level of Serum Procalcitonin prior to IV iron Infusion
Length of stay in the hospital | Up to 12 weeks
  Length of stay in the hospital
blood transfusions | Up to 12 weeks
  Number of blood transfusions
Diagnosis Related Groups (DRGs) related to infections | Up to 12 weeks
  Diagnoses encoding infections
Correlation of hepcidin and IV iron parameters | 4-28 days prior to elective surgery, IV iron is infused in the anesthesia pre-assessment clinic. Correlation of values prior to IV iron infusion, prior to surgery, at day 1, 3 and 7 or day of release from hospital
  Correlation of serum hepcidin and change of Hgb from baseline to day of surgery, day 1, 3 and 7 after surgery and the day of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Andrea U Steinbicker, Prof Dr MPH, Principal Investigator — Johann Wolfgang Goethe-University, Dept. of Anesthesiology, Intensive Care and Pain Medicine
Locations (2):
- Germany (2):
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - Dept. of Anesthesiology, Intensive Care and Pain Medicine, UKM, Münster

IPD SHARING:
Plan to Share IPD: No